CLINICAL TRIAL: NCT00841945
Title: Phase III Study of the Interest of Radiotherapy After 4 or 6 Cycles of CHOP 14 Rituximab Regimen of Chemotherapy , Patients With Agressive Localized Lymphoma
Brief Title: Treatment of Aggressive Localized Lymphoma
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: other drugs other studies
Sponsor: French Innovative Leukemia Organisation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GOELAMS 02 03
Record Dates: First submitted 2009-02-11; First posted 2009-02-12 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: B Cell Lymphoma
Keywords: Diffuse B larg cell lymphoma; Chemotherapy; Radiotherapy
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — Rituximab; Doxorubicin; Vincristine; Prednisone; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Chemotherapy + Radiotherapy
  - 4 or 6 R CHOP courses regimen every 14 days R CHOP = Rituximab, Doxorubicin, Vincristine and prednisone
  * Radiotherapy 40 gray on initial nodes
  Interventions: Drug: rituximab; Drug: doxorubicin; Drug: vincristine; Drug: prednisone; Procedure: radiotherapy
- 2 (Experimental): Chemotherapy
  - 4 or 6 R CHOP courses regimen every 14 days R CHOP = Rituximab, Doxorubicin, Vincristine and prednisone
  Interventions: Drug: rituximab; Drug: doxorubicin; Drug: vincristine; Drug: prednisone

INTERVENTIONS:
Drug: rituximab — RITUXIMAB 375 MG/M² IV DAY 1 or each course
  Other Names: MABTHERA
Drug: doxorubicin — doxorubicin 50 mg / m² iv day 1 of each course
  Other Names: Adriblastine
Drug: vincristine — VINCRISTINE 1?4 MG/M² IV ON DAY 1
  Other Names: Oncovin
Drug: prednisone — Prednisone 40 mg/m² DAy 1 to day 5
  Other Names: solupred
Procedure: radiotherapy — radiotherapy : total dose = 40 GY (5 fractions by week)
  Other Names: no other name
  Arms: 1

SUMMARY:
Prospective and multicentric Phase III study, evaluation of the interest of the radiotherapy after 4 or 6 cycles of CHOP 14 R regimen of chemotherapy , patients with agressive and localized B lymphoma , age 18 to 75 years.

DETAILED DESCRIPTION:
CHOP 14 R regimen of chemotherapy is a good standard in the treatment of agressive and localized B lymphoma.

Interest of the radiotheraphy

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 and < 75 years
* Diffuse B large cell lymphoma , CD 20+
* Ann Arbor stage I or II withe a bulk <7 cm
* stage i ou II confirmed by the PET-scan
* No previously treated
* HIV negative
* Signed Informed consent

Exclusion Criteria:

* Age< 18 and > 75 years
* other type of lymphoma
* CD20 negative
* Ann Arbor stage >II or bulk > 7 cm
* HIV positive
* Contraindication to Rituximab use according to Sm PC
* Containdication to antracyclin
* cancer or history of cancer , excepted in situ cancer of the cervix or skin epithelioma
* Refusal of sign the informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 334 (Actual)
Dates: Start 2005-04; Primary Completion 2016-01 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Event Free Survival (EFS) and Progression Free Survival (PFS) | EFS PFS one year after treatment

SECONDARY OUTCOMES:
Pet-scan | pronostic impact of Pet-scan
radiotherapy | Toxicity of the radiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Thierry LAMY, MD PhD, Principal Investigator — French Innovative Leukemia Organisation
Locations (1):
- Regional university hospital, Rennes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lamy T, Damaj G, Soubeyran P, Gyan E, Cartron G, Bouabdallah K, Gressin R, Cornillon J, Banos A, Le Du K, Benchalal M, Moles MP, Le Gouill S, Fleury J, Godmer P, Maisonneuve H, Deconinck E, Houot R, Laribi K, Marolleau JP, Tournilhac O, Branger B, Devillers A, Vuillez JP, Fest T, Colombat P, Costes V, Szablewski V, Bene MC, Delwail V; LYSA Group. R-CHOP 14 with or without radiotherapy in nonbulky limited-stage diffuse large B-cell lymphoma. Blood. 2018 Jan 11;131(2):174-181. doi: 10.1182/blood-2017-07-793984. Epub 2017 Oct 23. PMID 29061568
- [Derived] Tout M, Casasnovas O, Meignan M, Lamy T, Morschhauser F, Salles G, Gyan E, Haioun C, Mercier M, Feugier P, Boussetta S, Paintaud G, Ternant D, Cartron G. Rituximab exposure is influenced by baseline metabolic tumor volume and predicts outcome of DLBCL patients: a Lymphoma Study Association report. Blood. 2017 May 11;129(19):2616-2623. doi: 10.1182/blood-2016-10-744292. Epub 2017 Mar 1. PMID 28251914
- See also: FILO website — http://www.filo-leucemie.org